CLINICAL TRIAL: NCT06253260
Title: Analgesic Efficacy of Sequential Rapid Intrathecal Injection Of Dexmedetomidine Followed by Slow Injection of Hyperbaric Bupivacaine Versus Sequential Slow Injection of Both Drugs in Patients Undergoing Unilateral Inguinal Hernia Repair Surgery
Brief Title: Analgesic Efficacy of Sequential Rapid Versus Slow Intrathecal Injection Of Dexmedetomidine Followed by of Hyperbaric Bupivacaine in Inguinal Hernia Repair Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Omar Ahmed, Associate professor of Anesthesia, pain management & surgical ICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-367-2021
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Group A): rapid sequential group (Active Comparator)
  Interventions: Drug: Analgesic Efficacy of Sequential Rapid Intrathecal Injection Of Dexmedetomidine Followed by Slow Injection of Hyperbaric Bupivacaine Injection in Patients Undergoing Unilateral Inguinal Hernia Repair
- (Group B): normal sequential group (Active Comparator)
  Interventions: Drug: Analgesic Efficacy of Sequential Slow Intrathecal Injection Of Dexmedetomidine Followed by Slow Injection of Hyperbaric Bupivacaine in Patients Undergoing Unilateral Inguinal Hernia Repair Surgery

INTERVENTIONS:
Drug: Analgesic Efficacy of Sequential Rapid Intrathecal Injection Of Dexmedetomidine Followed by Slow Injection of Hyperbaric Bupivacaine Injection in Patients Undergoing Unilateral Inguinal Hernia Repair — Analgesic Efficacy of Sequential Rapid Intrathecal Injection Of Dexmedetomidine Followed by Slow Injection of Hyperbaric Bupivacaine Injection in Patients Undergoing Unilateral Inguinal Hernia Repair Surgery
  Arms: (Group A): rapid sequential group
Drug: Analgesic Efficacy of Sequential Slow Intrathecal Injection Of Dexmedetomidine Followed by Slow Injection of Hyperbaric Bupivacaine in Patients Undergoing Unilateral Inguinal Hernia Repair Surgery — Analgesic Efficacy of Sequential Slow Intrathecal Injection Of Dexmedetomidine Followed by Slow Injection of Hyperbaric Bupivacaine in Patients Undergoing Unilateral Inguinal Hernia Repair Surgery
  Arms: (Group B): normal sequential group

SUMMARY:
Analgesic Efficacy of Sequential Rapid Intrathecal Injection Of Dexmedetomidine Followed by Slow Injection of Hyperbaric Bupivacaine Versus Sequential Slow Injection of Both Drugs in Patients Undergoing Unilateral Inguinal Hernia Repair Surgery

DETAILED DESCRIPTION:
Once enrolled in the study, patients will be randomly assigned into two groups; rapid sequential group (Group A: n= 25) and normal sequential group (Group B: n=25). Randomization will be done by computer generated numbers and concealed by serially numbered, opaque and sealed envelopes. Upon arrival to the operating room, Wide bore intravenous line will be inserted, premedications (ondansetron 4 mg and midazolam 0.05 mg/Kg) will be administered, and routine monitors (Electrocardiogram - non-invasive blood pressure monitor - pulse oximeter) will be applied. The patient will be assisted into the sitting position, and sterilized surgical drapes will be placed to their back. Spinal anesthesia will be administered at L4-L5 using a complete aseptic technique. Group (A): will receive spinal anesthesia by applying sequential rapid injection of dexmedetomidine (5 µg in 0.5 ml saline, in insulin syringe within 1 second) followed by slow injection of 17.5 mg (3.5 ml within 12

-15 seconds) of 0.5% of heavy bupivacaine with no time lag between these injections. Group (B): will receive spinal anesthesia by applying normal sequential injection of 0.5 mL of 5 µg dexmedetomidine (injected over 3-4 seconds using a 5 ml syringe and mixed with cerebrospinal fluid (via barbotage), followed by slow injection of 17.5 mg (3.5 ml within 12 -15 seconds) of 0.5% of heavy bupivacaine with no time lag between these injections. Then the patient will be asked to lie down. The sensory level will be assessed by the cold ice technique every minute for 10-minutes. Motor blockade will be assessed every 5 min by the Bromage scale (4). After the T6 level is reached, the surgeon will be asked to operate. In case of failed spinal anesthesia (defined as failure to reach T6 level within 10 mins), the patient will be excluded, and further management will be according to the attending anesthetist. After spinal anaesthesia noninvasive blood pressure will be measured for then every 3 mins for 30 mins then every 5 mins till the end of operation. The occurrence of hypotension (defined as mean blood pressure <65 mmHg) will be recorded, and an anesthesiologist will be allowed to manage it by giving ephedrine (5-10 mg, intravenous [IV]) and IV fluids. If bradycardia occurred (heart rate<55 bpm), it will be managed by intravenous 0.5 mg atropine. Postoperative pain management All patients will receive acetaminophen 1gm/6 hours. Visual analogue scale (VAS) will be assessed at 0.5-, 1-, 2-, 4-, 6-, 8-, 10-, 12-,18- and 24-hour post operatively. Rescue analgesia administered in the form of (0.5-1 mg/kg) of intramuscular pethidine will be given on if VAS score was >3 Measurement tools

Patients will be monitored using:

* ECG, non-invasive blood pressure monitor, pulse oximeter.
* VAS (Visual analogue scale) pain assessment.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing inguinal hernia repair surgery.
* Age between 18 years and 65 years.
* Both sexes
* ASA I & ASA II

Exclusion Criteria:

* Patients refusal
* Pregnant women
* Duration of surgery more than 2 hours.
* Chronic use of opioids or tranquilizers.
* Incooperative patients e.g mentally retarded.
* Patients with any contraindications to spinal anesthesia
* Allergy to the used drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative analgesia | 24 hours
  time from reaching the sensory level of T6 until the need of first dose of rescue analgesia

SECONDARY OUTCOMES:
Onset of sensory block | 20 minutes
  defined as the time needed to lose cold sensation when using the ice-cold test at the T6 dermatomal level
Onset of motor block using Bromage scale | 30 minutes
  defined as the time from giving spinal anesthesia until a modified Bromage score of IV will be reached
VIisual Visual analouge scale Visual analogue scale (VAS) score at 0.5-, 1-, 2-, 4-, 6-, 8-, 10-, 12-, 18-and 24-hour post operatively | 24 hrs
  VAS score, a scale from 0 to 10, as 0 means no pain and 10 represents the most severe pain VAS score at 0.5-, 1-, 2-, 4-, 6-, 8-, 10-, 12-, 18-and 24-hour post operatively, a
Total dose of postoperative pethidine | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No